CLINICAL TRIAL: NCT00730873
Title: Fatty Liver and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Purpose: Treatment
Other Study IDs: 135/07
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obstructive Sleep Apnea
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

ARMS (1):
- A (Experimental): continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure

SUMMARY:
Non-alcoholic fatty liver disease is associated with obstructive sleep apnea. Abnormalities in liver enzymes can improve following continuous positive airway pressure in patients with obstructive sleep apnea. Computerized tomography can be used to quantify fatty liver changes. We hypothesize that continuous positive airway pressure can reduce morphologic fatty liver changes in patients with obstructive sleep apnea and non-alcoholic fatty liver, an that this reduction can be evident using computerized tomography

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea, defined as AHI>5/h

Exclusion Criteria:

* Consumption of more than 20 grams of alcohol per 24 h
* Known autoimmune disease
* Usage of known hepatotoxic drugs
* Medical history positive for viral hepatitis or other chronic liver disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Reduction in fatty liver changes on computerized tomography | Within 1-2 years

SECONDARY OUTCOMES:
Improved liver enzymes abnormalities | Within 1-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The pulmonary institute, Asaf Harofeh Medical Center, Ẕerifin, Israel